CLINICAL TRIAL: NCT05934474
Title: Biocollection on Peripheral Inflammation in Psychiatric Pathologies
Brief Title: Biocollection on Peripheral Inflammation
Acronym: IBIS-PSY
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: CR2TI, INSERM, UMR1064 (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC23_0270
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Schizoaffective Disorder, Depressive Type; Bipolar Disorder I; Bipolar Disorder II
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBIS-PSY patients
  Interventions: Biological: Peripheral venipuncture blood sampling, as part of standard care procedures; Other: Interview with a psychiatrist

INTERVENTIONS:
Biological: Peripheral venipuncture blood sampling, as part of standard care procedures — Collection of 36 mL of blood
Other: Interview with a psychiatrist — Research project data collection

SUMMARY:
Most psychiatric research is based on the nosographic classifications used in current practice. At present, there is no diagnostic or prognostic biomarker for psychiatric pathologies commonly used in clinical practice. The study hypothesis is that peripheral inflammatory biomarkers could be common to several psychiatric disorders, in particular psychotic disorders (bipolar disorder, schizophreniform disorder, schizophrenia, depressive episode with psychotic features). The aim of this project is to set up a bio-collection of biological samples (peripheral blood samples) with associated phenotypic data (assessment of various symptoms using standardized scales in patients whose blood is sampled). The setting up of this cohort follows on from work carried out on a PsyCourse cohort also using a transdiagnostic approach in psychiatry, in order to be able to collaborate within a European research project.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with one of the following diagnoses confirmed by a psychiatrist:

  * Characterized depressive episode with psychotic features,
  * Bipolar disorder type I
  * Bipolar disorder type II
  * Schizoaffective disorder
  * Schizophrenia
  * Schizophreniform disorder
* Patient under psychiatric care at Nantes University Hospital
* Patients weighing at least 45kg
* Patient affiliated to a social security scheme or beneficiary of such a scheme
* Patient who has given informed consent to participate in the study

Exclusion Criteria:

* Pregnant,
* History of cancer in the last 5 years,
* Vaccination within the last 4 weeks,
* Acute or chronic infection,
* Medical history of organ transplant,
* Medical history of autoimmune disease,
* Hearing impairment making it impossible to complete study questionnaires,
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited through the doctors who care for them on a regular medical basis, during a consultation or hospitalization in a psychiatric unit. After inclusion, an additional blood sample (4 tubes with a peripheral venous sample) will be taken by nurses from the psychiatric wards caring for the patient, during a blood sample taken as part of the patient's care. The sample will be transported to the Biological Resource Center (CRB) at Nantes University Hospital, where it will be stored along with all other study samples.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Demonstration of the presence of diagnostic biomarkers and biomarkers of severity common to several psychiatric disorders. | 2 hours
  Biological analysis of IBIS-PSY biocollection samples

SECONDARY OUTCOMES:
Validation of a patient clustering method separating patients with severe symptoms from those with mild symptoms | 2 hours
Replication of a pan-transcriptomic study (A Transcriptome-Wide Association Study (TWAS)) | 2 hours
Comparison of biomarkers between different psychiatric illnesses in order to develop models based on biological data that can help the physician adjust the diagnosis | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sauvaget, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No